CLINICAL TRIAL: NCT05001451
Title: A Phase 1, Open Label, Dose Escalation, and Dose Expansion Study to Assess the Safety, Tolerability, and Preliminary Antileukemic Activity of GDX012 in Patients With Minimal Residual Disease (MRD) Positive Acute Myeloid Leukemia
Brief Title: Study of GDX012 in Patients With MRD Positive AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This was a business decision to discontinue this clinical trial. The decision is not related to the safety of the investigational product, GDX012.
Sponsor: GammaDelta Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GDX012U-001
Record Dates: First submitted 2021-07-05; First posted 2021-08-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; MRD; gamma delta T-cells; allogeneic; cell therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GDX012 Suspension for IV Infusion (Experimental): Allogeneic cell therapy that is enriched for Vδ1+ γδ T cells
  Interventions: Biological: GDX012 Suspension for IV Infusion

INTERVENTIONS:
Biological: GDX012 Suspension for IV Infusion — Biological: GDX012 Suspension for IV Infusion (single dose) following chemotherapy for lymphodepletion.
  Drug: Fludarabine; chemotherapy for lymphodepletion
  Drug: Cyclophosphamide; chemotherapy for lymphodepletion

SUMMARY:
The purpose of this first-in-human study is to assess the safety, tolerability, antileukemic activity and maximum tolerated dose (MTD) of GDX012 in AML patients who are MRD positive by multiparametric flow cytometry.

The study will consist of a dose escalation stage to evaluate various doses of GDX012 after a lymphodepletion regimen comprising fludarabine and cyclophosphamide. Following determination of the MTD of GDX012, the study will expand at the MTD. Patients will be followed up for 12 months, after receiving GDX012.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Weight ≥ 40 kg
* Anticipated life expectancy > 3 months prior to lymphodepletion
* Karnofsky Performance Score ≥ 70%
* Histologically confirmed diagnosis of AML
* In complete response (CR) (including CRi/CRp); patients in first, second or subsequent CR (including CRi/CRp) are permitted
* MRD detected in bone marrow by MFC
* Negative pregnancy test (females of childbearing potential only)
* Agree to use effective birth control
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Platelet Count ≥ 20 x 109/L
* Prothrombin Time or INR ≤ 1.5 x ULN (unless receiving therapeutic anticoagulation)
* Partial Thromboplastin Time ≤ 1.5 x ULN (unless receiving therapeutic anticoagulation)
* Hemoglobin ≥ 8.0 g/dL
* Creatinine Clearance ≥ 40mL/min
* Serum Total Bilirubin ≤ 1.5 x ULN (unless documented Gilbert's Syndrome with Direct Bilirubin < 35% of Total Bilirubin)
* ALT ≤ 2.5 x ULN

Exclusion Criteria:

* Cytotoxic chemotherapy within 3 weeks
* Immune therapy within 4 weeks
* Immunosuppressive therapy within 2 weeks (with exceptions)
* Investigational treatment or interventional clinical trial within 4 weeks or 5 half-lives (if known), whichever is longer
* Major surgery within 4 weeks and/or not fully recovered from surgery-related toxicities
* Known hypersensitivity to chemotherapy, other agents, or excipients used in this study
* Female patient that is pregnant or lactating/breastfeeding
* Ongoing toxicity from prior anti-cancer therapy that have not recovered to ≤ Grade 1 (with exceptions)
* History of chronic or recurrent autoimmune or immune-mediated disease requiring steroids or other immunosuppressive treatments (including anti-tumor necrosis factor agents)
* Active CNS involvement (i.e. leukemic infiltration)
* Any other malignancy that requires active therapy
* Uncontrolled intercurrent illness (i.e. acute coronary syndrome in the last 6 months)
* Active infection with HIV, Hepatitis B or Hepatitis C

NOTE: other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (AEs) and serious adverse events (SAEs) | Up to 100 days
  AEs and SAEs occurring following administration of GDX012
Incidence of treatment emergent clinically significant abnormal laboratory assessments | Up to 100 days
  Standard clinical laboratory assessments for organ function (i.e. heart, kidney, liver)
Incidence of dose limiting toxicities (DLTs) | Up to 100 days
  DLTs occurring following administration of GDX012, measured using CTCAE 5.0 criteria
Establish the maximum tolerated dose (MTD) of GDX012 | Up to 100 days

SECONDARY OUTCOMES:
Evaluate the antileukemic activity of GDX012 | Up to 1 year
  Minimal residual disease (MRD) assessed by flow cytometry
Evaluate the antileukemic activity of GDX012 | Up to 1 year
  Incidence of patients converting from MRD positive to MRD negative
Evaluate the antileukemic activity of GDX012 | Up to 1 year
  Progression-free survival (PFS) and overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koslowski, MD, Study Director — GammaDelta Therapeutics Limited
Locations (1):
- City of Hope, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No